CLINICAL TRIAL: NCT04318223
Title: Palbociclib Plus Fulvestrant in Women With Hormone Receptor Positive and Human Epidermal Growth Factor Receptor Type 2 Negative Locally Advanced or Metastatic Breast Cancer Previously Treated With a CDK4/6 Inhibitor in Combination With Hormonal Therapy: a Multicenter, Phase II Trial
Brief Title: Palbociclib Plus Fulvestrant in Women With Hormone Receptor Positive and Human Epidermal Growth Factor Receptor Type 2 Negative Locally Advanced or Metastatic Breast Cancer Previously Treated With a CDK4/6 Inhibitor in Combination With Hormonal Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIM24-PALBO-BP
Record Dates: First submitted 2019-12-02; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer
Keywords: hormone receptor positive; human epidermal growth factor receptor type 2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: This is a Phase II, multicentre, single-arm study following a Simon's two-stage optimal design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm study following a Simon's two-stage optimal design (Experimental): Single-arm study with the primary objective of assessing the efficacy and safety of palbociclib in combination with fulvestrant (Faslodex) in women with HR+, HER2-negative metastatic breast cancer, regardless of their menopausal status, whose disease has progressed after prior treatment with AI plus a CDK4/6 inhibitor.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Patients will be enrolled into the study and assign to receive Palbociclib 125 mg/day orally for 3 weeks followed by 1 week off plus fulvestrant 500 mg intramuscularly on Days 1 and 15 of Cycle 1, every 28 days (+/- 7 days) thereafter starting from Day 1 of Cycle 1

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of palbociclib plus fulvestrant after failure of a combined treatment of hormonal therapy (aromatase inhibitor or tamoxifen ± LHRHa) plus a CDK4/6 inhibitor, in women with HR+ and HER2- LABC or MBC.

Primary endpoint:

1. To assess the clinical benefit rate (CBR) of the combination treatment palbociclib plus fulvestrant at progression of a combined treatment of hormonal therapy (aromatase inhibitor or tamoxifen ± LHRHa) and a CDK4/6 inhibitor.

   Clinical benefit rate for primary efficacy endpoints derivation will be based on the local (treating center's) radiologist's/investigator's tumor assessment.
   * For patients with measurable disease at baseline, progression will be determined according to the RECIST criteria v1.1.
   * In the absence of measurable disease at baseline, patients with bone only lesions, lytic or mixed (lytic + sclerotic), will be allowed to enter the study and the following will be considered disease progression among these patients:
   * The appearance of one or more new lytic lesions in bone,
   * The appearance of one or more new lesions outside of bone,
   * Unequivocal progression of existing bone lesions.

   Note: Pathologic fracture, new compression fracture, or complications of bone metastases will not be considered as evidence of disease progression, unless one of the above-mentioned criteria is fulfilled.
2. To assess the Quality of Life (QoL) of patients receiving the combination treatment palbociclib plus fulvestrant at progression of a combined treatment of hormonal therapy (aromatase inhibitor or tamoxifen ± LHRHa) and a CDK4/6 inhibitor.

Secondary Endpoints:

1. To evaluate the efficacy of the combination of fulvestrant plus palbociclib at the progression of a combined treatment of hormonal therapy (aromatase inhibitor or tamoxifen ± LHRHa) and CDK4/6 inhibitors with respect to:

   * Overall response rate (ORR)
   * Progression Free Survival (PFS)
   * Overall Survival (OS)
   * Safety and tolerability
2. To assess predictive biomarkers of response/resistance to fulvestrant plus palbociclib using metastatic tumor tissue samples and liquid biopsies.

This study will be performed in pre- and post-menopausal women with HR+/HER2- LABC or MBC whose disease is progressing to a CDK4/6 inhibitor in combination with hormonal therapy (aromatase inhibitor or tamoxifen ± LHRHa).

Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first.

DETAILED DESCRIPTION:
This is a Phase II, multicentre, single-arm study following a Simon's two-stage optimal design

Screening phase At screening, the investigator or his/her authorized designee will assign a unique number to patients being considered for the study. The patient should provide a signed Informed Consent Form prior to any study screening evaluations. Once the patient Informed Consent Form has been signed and eligibility is confirmed (all inclusion/exclusion criteria has been verified), the patient can be enrolled. All screening evaluations will be performed within 28 days prior to Treatment Day 1. Patients may be re-screened.

Treatment phase Eligible patients will receive Fulvestrant plus palbociclib. Patients will be treated with fulvestrant 500 mg i.m. on Days 1, 15 and 29 and every 28 days thereafter and palbociclib125 mg oral day 1 to 21 every 28 days.

Dose adjustment (reduction, interruption) according to toxicity of study treatment will be allowed. Study treatment will continue until one of the following conditions apply - whichever comes first:

* tumor progression
* unacceptable toxicity according to investigator's judgment
* death
* discontinuation from the study for any other reason Further treatments after discontinuation will be at the investigator's discretion. During the study, visits will be performed monthly and at the end of treatment. Tumor assessment will be performed every 3 cycle of treatment.

For each patient enrolled in the present study a blood sample (mandatory) at study enrollment and at disease progression (mandatory) will be provided. Additionally, a tissue sample from the most accessible metastatic site will be collected at study enrollment and at disease progression (optional). Blood and tumor samples will be used to investigate the mechanisms of response and resistance to therapy with palbociclib in combination with fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years of age) pre or post-menopausal women with LABC or MBC not amenable to curative treatment by surgery or radiotherapy, progressing to a CDK4/6 inhibitor in combination with aromatase inhibitor or tamoxifen in the adjuvant or metastatic setting. To be enrolled in the present trial patients must have relapsed at least after 12 months from the last CDK4/6 dosage in the adjuvant setting or at progression from a first line combined hormonal treatment for metastatic disease with a CDK4/6 inhibitor plus AI or Tam with duration of, at least, 6 months. For metastatic disease, patients must have achieved, at least a stable disease while the first line hormonal treatment with a CDK4/6 inhibitor plus AI or Tam to be enrolled in the trial.
2. Patients receiving up to one line of chemotherapy before the first line hormonal treatment with a CDK4/6 inhibitor for metastatic disease may be enrolled in the study.
3. Histological confirmation of ER and/or PgR ≥ 1% and HER2 negative breast cancer (IHC status 0, 1+, 2+ and FISH not amplified).
4. Premenopausal women: in order to be eligible must have achieved surgical menopause with bilateral oophorectomy or ovarian radiation or medical menopause by treatment with a luteinizing hormone-releasing hormone (LHRH) agonist (LHRHa) for induction of ovarian suppression.
5. Radiological or objective evidence of recurrence or progression on or after the last systemic therapy prior to enrollment.
6. Patients who received ≤ 28 days of fulvestrant for second line advanced breast cancer treatment prior to study enrollment are eligible.
7. Patients must have:

   * At least one lesion that can be accurately measured in at least one dimension ≥ 20 mm with conventional imaging techniques or ≥ 10 mm with spiral CT or MRI
   * Bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease as defined above.
8. Adequate bone marrow and coagulation and adequate organ function defined as follows:

   * ANC > 1,000/mm3 (1.0 x 109/L);
   * Platelets > 75,000/mm3 (75 x 109/L);
   * Hemoglobin≥ 9 g/dL (90 g/L);
   * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution;
   * Total serum bilirubin≤1.5 x ULN (<2.5 ULN if Gilbert's disease);
   * AST and/or ALT≤ 3 x ULN (≤ 5 x ULN if liver metastases present);
   * Alkaline phosphatase ≤2.5 x ULN (≤ 5 x ULN if bone or liver metastases present);
   * ECOG Performance Status≤ 2;
   * Resolution of all acute toxic effects of prior therapy or surgical procedures to National Cancer Institute (NCI) CTCAE Grade ≤1 (except alopecia).
9. Estimated life expectancy of >12 weeks.
10. Patients must perform liquid biopsy at study entry and at disease progression. Tissue biopsy of the most accessible metastatic site at study entry and at disease progression are required but not mandatory.
11. Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion Criteria:

1. HER2-overexpressing patients by local laboratory testing (IHC3+ staining or in situ hybridization positive).
2. Patients who received > 1 line of chemotherapy as treatment for MBC.
3. Patients who received > 1 line of a CDK4/6 inhibitor in combination with hormonal treatment for LABC or MBC or who have relapsed at less than 12 months from the end of adjuvant treatment with a CDK4/6 inhibitor. For metastatic disease, patients with a progressive disease within the first 6 months of treatment while on first line therapy with a CDK4/6 inhibitor, will be excluded.
4. Patients receiving chemotherapy or any type of hormonal therapy after treatment with a CDK4/6 inhibitor for metastatic disease.
5. Patients interrupting the previous treatment with CDK4/6 inhibitor for cardiac and/or hepatic toxicity and not for disease progression.
6. Pregnant, lactating women.
7. Known hypersensitivity to CDK4/6 inhibitors, fulvestrant, or to any of the excipients.
8. Radiotherapy within four weeks prior to enrollment (baseline/treatment start) except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to enrollment (baseline/treatment start). Patients must have recovered from radiotherapy toxicities prior to enrollment.
9. Currently receiving hormone replacement therapy, unless discontinued prior to enrollment.
10. Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use, at the time of study entry except in cases outlined below:

    1. short duration (<2 weeks) of systemic corticosteroids is allowed (e.g., chronic obstructive pulmonary disease, anti-emetic);
    2. low doses of corticosteroids for brain metastasis treatment is allowed.
11. Patients with symptomatic visceral disease in need of urgent disease control (e.g., significant dyspnea related to pulmonary lymphangitic carcinomatosis and lung metastases or clinically meaningful symptomatic liver metastasis at the judgement of treating investigator).
12. Symptomatic brain metastases.
13. Patients with a known history of HIV seropositivity.
14. Active, bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin, low-molecular-weight heparin (LMWH) and acetylsalicylic acid or equivalent, as long as the INR is ≤ 2.0).
15. Any severe and/or uncontrolled medical conditions such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to enrollment, serious uncontrolled cardiac arrhythmia.
16. Acute and chronic, active infectious disorders.
17. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study treatments (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome).
18. Inability to swallow oral medications.
19. Significant symptomatic deterioration of lung function.
20. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itroconazole, Voriconazole, Ritinavir, Telithromycin) within the last 5 days prior to enrollment.
21. History of non-compliance to medical regimens.
22. Patients refusing to perform liquid biopsy at study entry and disease progression.
23. Patients unwilling to or unable to comply with the protocol.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Response (CBR) | About 48 months
  To assess the clinical benefit rate (CBR) of the treatment, the Clinical Benefit Response (CBR) is defined as complete response (CR) or partial response (PR) or stable disease (SD) >24 weeks according to the RECIST version 1.1 recorded in the time period between enrollment and disease progression or death of any cause. CBR with the corresponding 95% Confidence Interval (95% C.I.) will be estimated using the exact binomial method. A Simon optimal two-stage design will be used to exclude a clinical benefit rate (CBR) of 30% (p0 = 0.30) with a clinical relevant target of 40% (p1 = 0.40) using a one-sided alpha-level of 0.05 and a power of 0.80. Fifty-nine (59) subjects will be enrolled in the first phase. If nineteen (19) of fewer CR+PR+SD will be observed, the study will be terminated. Otherwise the treatment will be considered worthy of further investigation and 109 more subjects will be enrolled for a total sample size of 168 subjects.
Patient Reported Outcomes (PRO) | About 48 months
  Breast cancer-specific quality of life total scale scores and single item scale scores will be summarized by descriptive summary tables at baseline and over time. The mean changes from baseline will also be summarized using descriptive statistics. Longitudinal trajectories of total scale scores will be modelled using linear mixed models with random intercept to account for subject specific baseline assessment; time will be modeled continuously using days since baseline; potential non linear trend will be examined by adding quadratic terms to the model. Selection of the best model will be based on Akaike Information Criterion (AIC).

SECONDARY OUTCOMES:
Efficacy of the combination of fulvestrant plus palbociclib | About 48 months
  To evaluate the efficacy of the combination of fulvestrant plus palbociclib at the progression of a combined treatment of hormonal therapy and CDK4/6 inhibitors with respect to:
  • Overall response rate (ORR) :will be estimated by dividing the number of patients with OR (CR or PR) by the number of patients ("response rate"). A 95% CI for the response rates will be provided using the exact binomial method
Efficacy of the combination of fulvestrant plus palbociclib | About 48 months
  To evaluate the efficacy of the combination of fulvestrant plus palbociclib at the progression of a combined treatment of hormonal therapy and CDK4/6 inhibitors with respect to:
  • Overall Survival (OS) :the median event times and 95% CIs will be estimated. The 1-year survival probability will be estimated using the Kaplan-Meier method and a two sided 95% CI for the log [-log(1-year survival probability)] will be calculated using a normal approximation using the Greenwood's formula
Efficacy of the combination of fulvestrant plus palbociclib | About 48 months
  To evaluate the efficacy of the combination of fulvestrant plus palbociclib at the progression of a combined treatment of hormonal therapy and CDK4/6 inhibitors with respect to:
  • Progression Free Survival (PFS) :the analyses of PFS will be performed in the ITT population. PFS time will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. 95% CIs for the 25th, 50th and 75th percentiles of the event-free time (if reached) will be reported.
Predictive biomarkers of response/resistance | About 48 months
  To assess predictive biomarkers of response/resistance to fulvestrant plus palbociclib using metastatic tumor tissue samples and liquid biopsies. Patients must perform liquid biopsy at study entry and at disease progression.
  Biopsies will be used to investigate expression levels and/or genetic alteration of cell cycle components as well as additional molecular pathways potentially responsible for resistance to CDK4/6 inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine De Angelis, MD, Study Director — Federico II University
Locations (19):
- Italy (19):
  - Nuovo ospedale di Prato - S. Stefano, Prato, Firenze
  - Ospedale Civile S. Giovanni di Dio, Frattamaggiore, Napoli
  - Centro di Riferimento oncologico, Aviano, Pordenone
  - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Ospedale Sacro Cuore di Gesù Fatebenefratelli, Benevento
  - A.O. Osp. Riuniti - ASST PAPA GIOVANNI 23, Bergamo
  - Ospedale di Brindisi "Perrino", Brindisi
  - Ospedale Policnico San Martino, Genova
  - Ospedale Vito Fazzi, Lecce
  - Azienda Ospedaliera Papardo, Messina
  - Azienda Ospedaliero - Universitaria di Modena, Modena
  - A.O.U. Seconda Universita' degli Studi di Napoli, Napoli
  - Azienda Ospedaliera 'A. CARDARELLI', Napoli
  - Azienda Ospedaliera dei Colli - P.Monaldi, Napoli
  - Istituto Nazionale Tumori IRCCS Pascale, Napoli
  - Università degli Studi di Napoli "Federico II", Napoli
  - A.O.U. Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena (IRE, Roma
  - Ospedale Sandro Pertini, Roma